CLINICAL TRIAL: NCT03370107
Title: Comparison of the Analgesic Effects of Two Methods of Repetitive Magnetic Transcranial Stimulation: A Randomized Double Blind Sham Controlled Study in Patients With Central Neuropathic Pain
Brief Title: Comparison of rTMS and H Coil in Neuropathic Pain
Acronym: HNEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Nadine ATTAL, Principal investigator and coordinator, Hospital Ambroise Paré Paris
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HNEP4
Record Dates: First submitted 2017-12-01; First posted 2017-12-12 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Central Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of 2 treatment groups: active rTMS and Hcoil or sham rTMS and sham Hcoil, according to a 2 : 1 ratio (2 for active, 1 for placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The sham coil of the Hcoil procedure produces a similar acoustic artefact and scalp sensation as the active coil and mimics the facial muscle activation induced by the active coil. The sham stimulation of the conventional rTMS will be carried out with the opposite face of the coil (biface coil) of identical size, color and shape emitting a sound similar to that emitted by the active coil (B65 A/P Butterfly Coil Magventure).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS and H coil (Active Comparator)
  Interventions: Device: rTMS
- sham rTMS and Hcoil (Placebo Comparator)
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Conventional magnetic stimulations will be applied with a MacPROX100 machine using neuronavigation system. H-coil rTMS will be delivered with the Brainsway H-coil (Brainsway, Jerusalem, Israel) applied via a helmet placed on the head corresponding to the primary motor cortex (H10 coil) and connected to a Masgtim Rapid2 stimulatior (Mastim, Whitland, UK), while sham stimulation will be delivered with a sham coil placed in the helmet encasing the active rTMS coil. Active rTMS sessions with H-coil will use exactly the same parameters of stimulation as conventional rTMS.

SUMMARY:
rTMS of the motor cortex is an increasingly established analgesic technique for the treatment of neuropathic pain. However its efficacy is generally modest. One reason may be the that conventional rTMS targets only superficial and small cortical regions of the human brain. A newer cooled coil, the Hesed (H) coils, now allows deep and larger surface of stimulation and has been suggested to have analgesic effects in a small pilot trial in diabetic painful polyneuropathy. Based on its deeper mechanism of action and larger surface of stimulation, we hypothesize that this technique will be more effective than rTMS in patients with central pain, a highly unmet medical need. The primary objective of the present study will be to compare the efficacy of H coil, conventional rTMS and sham stimulation of the primary motor cortex in patients central neuropathic pain. Major secondary objectives will be to directly compare the analgesic efficacy of H coil versus conventional rTMS, and compare the efficacy of both techniques in patients with lower limb pain and those with upper limb pain/face. This will be a randomized tricentric sham controlled study

DETAILED DESCRIPTION:
This will be a tricenter randomized double blind sham controlled trial with stratified randomization based on the area of pain. Patients will first undergo MRI of the skull to determine the exact position of the coil of the motor cortex for neuronavigation with conventional rTMS. After providing informed consent, they will be randomly assigned to one of 2 treatment groups: active rTMS and Hcoil or sham rTMS and sham Hcoil, according to a 2 : 1 ratio (2 for active, 1 for placebo). For each treatment group (active or sham), the order of sessions will be again randomized according to a crossover design : thus each patient will receive successively either active rTMS followed by active H coil or active H coil followed by active rTMS or two sham stimulations (rTMS and H coil). Each treatment will be applied by an independent investigator not involved in the assessment or selection of patients. The treatment protocol will include 2 periods separated by an interval of 5 to 6 weeks depending on the potential residual analgesic effects to avoid carryover effects (patients whose pain intensity remains minimal after 6 weeks, eg less than 4 /10 on NRS, will not participate in the second crossover period of the study). Each session will consist of 5 consecutive stimulation visits of (active or sham) rTMS and H coil over 5 consecutive days. Each patient will thus receive a total of 10 stimulations (2 series of 5 active rTMS or H coil or 2 series of 5 sham rTMS or H coils) and will have a total of 15 visits, including one screening visit (V1), 10 stimulation visits (V2-V5 and V8-V13), and 4 poststimulation visits 1 and 3 weeks after each treatment period (V6, V7, V14, V15). Conventional magnetic stimulations will be applied with a MacPROX100 machine using neuronavigation system and sessions will consist of 30 series of 10 second pulses with a frequency of 10 Hz and an interval of 20 seconds between each. The stimulation intensity used will be 80 % of the resting motor threshold. Conventional rTMS stimulations will target the primary motor cortex contralateral to the painful area or left side in case of bilateral pain and sham stimulation will be carried out with the opposite face of the coil (biface coil) of identical size, color and shape emitting a sound similar to that emitted by the active coil. H-coil rTMS will be delivered with the Brainsway H-coil (Brainsway, Jerusalem, Israel) applied via a helmet placed on the head corresponding to the primary motor cortex (H10 coil) and connected to a Masgtim Rapid2 stimulatior (Mastim, Whitland, UK), while sham stimulation will be delivered with a sham coil placed in the helmet encasing the active rTMS coil. Active rTMS sessions with H-coil will use exactly the same parameters of stimulation as conventional rTMS, e.g. 30 consecutive trains of stimuli delivered at 10 Hz, at 80 % resting motor threshold (RMT), separated by intertrain intervals of 20 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years and less than 80 years
* Average pain intensity ≥ 4/10 at screening and randomization
* Persistent pain for at least 6 months
* Stable pharmacological treatment for pain
* Central neuropathic pain as diagnosed by DN4 and NeuPSIG classification algorithm related to stable multiple sclerosis, spinal cord lesion or past stroke

Exclusion Criteria:

* Any clinically significant or unstable medical or psychiatric disorder
* History of substance abuse
* Litigation
* Pregnancy/lactation
* Contraindication to rTMS or Hcoil
* Intermittent pain, more severe pain than neuropathic pain and diffuse pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change in the self reported average pain intensity (NRS from 0 to 10) over the past 24 hours from baseline to week 3 after the end of the last stimulation | the average of pain scores (NRS for pain intensity) will be conducted before each treatment for up to 3 weeks after each treatment session (treatment effect)
  Comparison between the efficacy of sham, rTMS and H coil on average pain intensity over the course of the treatment

SECONDARY OUTCOMES:
Score of each neuropathic dimension (ie symptom combinations) on the Neuropathic pain symptom inventory (NPSI) (Bouhassira et al 2004) . | 1 week and 3 weeks after the end of each stimulation period
  This validated questionnaire for neuropathic pain quantifies the mean intensity of 10 neuropathic symptoms and their combination into 5 distinct dimensions during the last 24 hours on 11-point (0-10) numerical scales.
proportion of responders | 1 week and 3 weeks after the end of each stimulation period
  proportion of patients achieving at least 30 % and 50 % pain relief as compared to prestimulation values allowing to calculate Numbers Needed to Treat for 30 % and 50 % pain relief.
intensity of average pain | 1 week and 3 weeks after the end of each stimulation period
  Numerical pain scale for average pain intensity from the the Brief Pain Inventory (BPI) rated from 0 (no pain) to 10 (maximal pain imaginable)
Pain interference | 1 week and 3 weeks after the end of each stimulation period
  7 items for pain interference of the BPI rated from 0 (does not interfere), to 10 (complete interference) to measure the impact of pain on general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life
Hospital Anxiety and Depression Scale (HAD) | 1 week and 3 weeks after the end of each stimulation period
  14 items scored as anxiety and depression scores (each on 21)
French version of the Pain Catastrophizing Scale (PCS) | 1 week and 3 weeks after the end of each stimulation period
  The PCS consists of 13 items describing the thoughts and feelings that individuals may experience when in pain (range 0-52); the patients' overall impression of change (PGIC) on a 7-point scale (from very much improved to very much worse).
Intensity of maximal pain over the past 24 hours | 1 week and 3 weeks after the end of each stimulation period
  Maximal pain intensity from the Brief Pain Inventory
sensory and affective score of the short form McGill Pain questionnaire | 1 week and 3 weeks after the end of each stimulation period
  15 items, of which 11 assess the sensory dimension of pain (rated on 44) and 4 assess the affective dimension of pain (rated on 15).
Intensity of least pain over the past 24 hours | 1 week and 3 weeks after the end of each stimulation period
  Intensity of least pain on NRS from the Brief Pain Inventory
intensity of brush induced allodynia | 1 week and 3 weeks after the end of each stimulation period
  measured with a brush (SOMEDIC) (mean of 3 stimulations) in the area of maximal pain on a 0-10 NRS
side effects | immediately after each rTMS session
  specific side effects questionnaire specifically designed for assessment of safety in rTMS studies
blinding | 3 weeks after the end of the second stimulation period
  blinding questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nadine ATTAL, Study Director — Coordinator of the study
Locations (1):
- Department of Pain Management and Research, Oslo University Hospital and Faculty of Medicine, University of Oslo, Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
No plan to make individual participant data available to other researchers